CLINICAL TRIAL: NCT03602170
Title: Cardiovascular Effects of High-Intensity Interval Training (HIIT) and Moderate-Intensity Continuous Training (MCT)
Brief Title: Cardiovascular Effects of High-Intensity Interval Training (HIIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, David Edwards, Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1009103-6
Record Dates: First submitted 2018-06-21; First posted 2018-07-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Healthy Sedentary Adults With BP <140/90
Keywords: High-Intensity Interval Training; Exercise; Cardiovascular Health; Blood Pressure
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Interval Training (Experimental): 8 weeks of high-intensity interval training. Three sessions per week will be performed (24 total sessions).
  Interventions: Behavioral: High-Intensity Interval Training
- Moderate-Intensity Continuous Training (Active Comparator): 8 weeks of moderate-intensity continuous training. Three sessions per week will be performed (24 total sessions).
  Interventions: Behavioral: Moderate-Intensity Continuous Training

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — Supervised exercise sessions will be performed on a upright cycle ergometer. Training sessions involve 20 minutes of exercise by completing 10 repetitions of 60 seconds of exercise at 90-95% maximal heart rate with 60 seconds of active rest between each repetition at 50-60% maximal heart rate.
  Arms: High-Intensity Interval Training
Behavioral: Moderate-Intensity Continuous Training — Supervised exercise sessions will be performed on a upright cycle ergometer. Training sessions involve 30 minutes of continuous exercise at 65-70% maximal heart rate.
  Arms: Moderate-Intensity Continuous Training

SUMMARY:
The purpose of this study is to determine the effect of high-intensity interval training (HIIT) in comparison to moderate-intensity continuous training (MCT) on blood pressure, blood vessel function, and blood pressure reactivity.

DETAILED DESCRIPTION:
It is estimated that one-third of the adult population in the United States has blood pressure values that are classified as prehypertension. This slight elevation in blood pressure has been shown to result in an increased risk for developing hypertension and cardiovascular disease. The Seventh Report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure (JNC7) recommends lifestyle modifications for individuals classified as prehypertensive. One lifestyle modification suggested by JNC7 is regular physical activity. Aerobic exercise, like moderate-intensity continuous training (MCT), has been shown to improve blood pressure, blood vessel function, and arterial stiffness in those with prehypertension. However, a major barrier to exercise adherence is the time commitment required. High-Intensity Interval Training (HIIT), which requires individuals to work at higher intensities for shorter durations, may offer an alternative training design that would reduce the time commitment. Previous studies have shown HIIT to be equal to or better at improving cardiorespiratory fitness and blood vessel function in multiple populations. Limited information is present on HIIT training in those with prehypertension. In this study, participants will be randomized into one of the two training program designs mentioned above (MCT or HIIT). Both programs will be completed over an 8-week period (3 sessions per week) and each training session will be supervised. Participants will complete testing visits before and after the training program to collect measures of cardiovascular health (exercise capacity, blood pressure, blood vessel function, and blood pressure reactivity). The goal is to compare the effects of the training programs on these measures of cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Blood Pressure less than 140/90 mmHg
* Sedentary

Exclusion Criteria:

* Known or major signs/symptoms of cardiovascular, pulmonary, renal, or metabolic disease
* Cancer
* Use of antihypertensive medication
* Current tobacco use
* BMI (body mass index) less than 30 kg/m2
* Postmenopausal
* Current pregnancy
* Current hormone replacement therapy
* Participating in regular aerobic exercise at least three times a week for 30 minutes at a moderate intensity for the past 3 months or more
* Not able to regularly exercise for any reason

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Change from baseline resting blood pressure at 8 weeks
  Resting blood pressures measuring by automated oscillometric device

SECONDARY OUTCOMES:
Peak Aerobic Capacity | Change from baseline VO2peak at 8 weeks
  Peak oxygen uptake (VO2peak/max) during incremental cycling exercise until exhaustion
24-Hour Ambulatory Blood Pressure | Change from baseline 24-hour ambulatory blood pressure at 8 weeks
  24 hours of continuous ambulatory blood pressure monitoring by oscillometric device
Pulse Wave Analysis | Change from baseline central blood pressure measures at 8 weeks
  Central blood pressure measures assessed by radial tonometry
Endothelial Function | Change from baseline endothelial function at 8 weeks
  Assessed by brachial artery flow mediated dilation and change in blood in femoral artery in response to passive limb movement
Arterial stiffness | Change from baseline pulse wave velocity measures at 8 weeks
  Pulse wave velocity measures (carotid to femoral and femoral to distal) assessed by applanation tonometry
Blood Pressure Reactivity | Change from baseline blood pressure reactivity at 8 weeks
  Blood pressure response to graded exercise test and handgrip exercise

OTHER OUTCOMES:
Perceived Enjoyment of Exercise | Measured after 4 and 8 weeks of training
  Enjoyment rating based on 18-item questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Bryce J Muth, MS, Principal Investigator — University of Delaware; David G Edwards, PhD, Principal Investigator — University of Delaware
Locations (1):
- Department of Kinesiology and Applied Physiology, University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided